CLINICAL TRIAL: NCT00730743
Title: Open Liver Resection With or Without Vascular Inflow Occlusion: a Randomized Control Trial
Brief Title: Study on Clinical Outcome of Vascular Inflow Occlusion in Open Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yue Sun, Associate Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT08017; CRE-2008.037-T
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intermittent clamp group
  Interventions: Procedure: Intermittent Pringle maneuver
- 2 (No Intervention): No clamp group

INTERVENTIONS:
Procedure: Intermittent Pringle maneuver — Pringle maneuver is performed by isolation of the hepatoduodenal ligament which is then encircled and occluded with atraumatic vascular clamp. The clamp is applied for 15 minutes followed by unclamping for 5 minutes and repeated till end of liver transection. Limits of clamp cycle: 3 cycles for cirrhotic liver; 4 cycles for non-cirrhotic liver.
  Arms: 1

SUMMARY:
This study aims to evaluate whether applying inflow vascular occlusion in modern liver resection is associated with better clinical outcome.

Eligible patients are randomly assigned to the two surgical techniques: with or without the application of inflow vascular occlusion.

Patients outcome including liver function recovery, operative time and blood loss are compared.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Child-Pugh Class A or B

Exclusion Criteria:

* Informed consent not available
* Presence of portal vein thrombosis, portal vein tumor thrombus, or previous portal vein embolisation
* Presence of hepatic artery thrombosis, previous transarterial therapy like TACE, or transarterial internal radiation
* When portal vein resection is anticipated
* Emergency hepatectomy
* Ruptured hepatocellular carcinoma
* Rehepatectomy (repeated liver resection)
* Adhesion or anatomical variation that preclude safe and successful application of Pringle maneuver
* When concomitant bowel or bile duct resection is anticipated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Operative blood loss | From skin incision to completion of operation
Operative time | From skin incision to completion of operation

SECONDARY OUTCOMES:
Operative morbidity and mortality | From date of operation to 30-day after operation
Recovery of liver function | From date of operation to date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kit-fai Lee, MBBS, Principal Investigator — Departement of Surgery, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Lee KF, Chong CCN, Cheung SYS, Wong J, Fung AKY, Lok HT, Lai PBS. Impact of Intermittent Pringle Maneuver on Long-Term Survival After Hepatectomy for Hepatocellular Carcinoma: Result from Two Combined Randomized Controlled Trials. World J Surg. 2019 Dec;43(12):3101-3109. doi: 10.1007/s00268-019-05130-8. PMID 31420724
- [Derived] Lee KF, Cheung YS, Wong J, Chong CC, Wong JS, Lai PB. Randomized clinical trial of open hepatectomy with or without intermittent Pringle manoeuvre. Br J Surg. 2012 Sep;99(9):1203-9. doi: 10.1002/bjs.8863. Epub 2012 Jul 24. PMID 22828986